CLINICAL TRIAL: NCT01494896
Title: An Open-Label Study to Explore the Impact of Inhaled Treprostinil Sodium on Ventilation Perfusion Matching When Used for Treatment of Group 1 Pulmonary Arterial Hypertension in Patients With Concomitant Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Impact of Inhaled Treprostinil Sodium on Ventilation Perfusion Matching
Status: Terminated | Type: Observational
Why Stopped: due to slow enrollment. United Therapeutics and Dr. Bajwa MD decided to terminate study
Sponsor: University of Florida (Other)
Collaborators: United Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: Tyvaso COPD
Record Dates: First submitted 2011-12-15; First posted 2011-12-19 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2013-08

CONDITIONS: Pulmonary Arterial Hypertension; Chronic Obstructive Pulmonary Disease
Keywords: Pulmonary Hypertension; Pulmonary Arterial Hypertension; COPD; Chronic Obstructive Pulmonary Disease; Tyvaso; Inhaled Treprostinil Sodium; Ventilation Perfusion Matching; HO Group 1 Pulmonary Arterial Hypertension; Concomitant Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Pulmonary Disease, Chronic Obstructive; Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to see how inhaled treprostinil sodium (Tyvaso) affects the amount of air and blood that reach the alveoli, or tiy air sacs, in the lungs of patients with Group 1 Pulmonary Arterial Hypertension with concomitant Chronic Obstructive Pulmonary Disease (COPD).

DETAILED DESCRIPTION:
In patients with severe COPD where the FEV1 is 50% or less than predicted, emphysema and obliterating bronchiolitis presenting a "ceiling" to any improvement in function that can be achieved by therapies that dilate the airways or lessen inflammation. Such severe COPD is commonly associated with pulmonary hypertension at rest or during exercise. Although hypoxia has been classically considered to be the major pathogenic mechanism of pulmonary hypertension in COPD and oxygen has been the mainstay of therapy, other mechanisms may play important roles. Indeed, endothelial dysfunction can be observed in patients with mild to moderate COPD who do not have hypoxemia and in smokers with normal lung function. In addition, long-term oxygen therapy does not generally result in resolution of the pulmonary hypertension. A key question that remains is whether the newer therapies for pulmonary arterial hypertension (PAH) could improve pulmonary hypertension and therefore exercise tolerance in COPD.

Unfortunately the use of non-selective pulmonary vasodilator therapy in oral, intravenous or subcutaneous form for PAH patients who have unrelated concomitant COPD, is known to cause worsening gas exchange and intensification of symptoms despite a decrease in pulmonary vascular resistance and arterial pressures.

We hypothesize that an inhaled pulmonary vasodilator may not worsen ventilation-perfusion mismatching by selectively vasodilating well ventilated areas in PAH patients with concomitant COPD and in fact may improve ventilation perfusion matching leading to preservation or improvement of oxygenation.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a diagnosis of PAH confirmed by right heart catheterization within the last 12 months (defined by mean pulmonary artery pressure of greater than or equal to 25 with pulmonary capillary wedge pressure or left ventricular end-diastolic pressure of less than or equal to 15).
* Subject is being initiated on inhaled treprostinil for treatment of PAH.
* Subject between 18 and 80 years of age at screening with a diagnosis of COPD confirmed by spirometry within the last 6 months showing FEV1 > 40% predicted and FEV/FVC of < 70.
* Baseline 6-minute walk distance > 150 meters.
* Subject has not been on any approved therapy for their PH for the last 90 days.
* If subject is being treated with conventional therapy for COPD, they must be receiving a fixed regimen of these therapies for tat least 30 days prior to Baseline.
* Previous echocardiography with evidence of normal left systolic and diastolic ventricular function, and absence of any clinically significant left sided heart disease.
* If female, physiologically incapable of childbearing or practicing an acceptable method of birth control as deemed appropriate by the physician or institution.
* If female, negative serum pregnancy test required at screening.
* Subject voluntarily gives informed consent.

Exclusion Criteria:

* The subject is pregnant or lactating.
* Subject has had a new type of chronic therapy for PH added within 90 days of Baseline.
* Subject has had any medication started or discontinued for COPD within 30 days of Baseline.
* Subject has any of the following: portal hypertension, chronic thromboembolic disease, pulmonary veno-occlusive disease or other than those accepted as part of the inclusion criteria or has had any atrial septostomy.
* Subject has a current diagnosis of uncontrolled sleep apnea as defined by their physician.
* Subject has a history or current evidence of left-sided heart disease.
* Subject has interstitial lung disease as evidence by CT scan or restrictive pattern on pulmonary function tests (FEV1/FVC > 70 and TLC < 80% predicted) or COPD with FEV1 < 40% predicted.
* Subject has a musculoskeletal disorder or any other disease that is likely to limit ambulation, or is connected to a machine that is not portable.
* Subject is incapable of maintaining compliance throughout the course of the study.
* Any condition, in the investigator's opinion, would constitute an unacceptable risk to the subject's safety.
* Subject is receiving an investigational drug, has an investigational device in place or has participated in an investigational drug or device study within 30 days prior to screening.
* Subjects without a telephone contact.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects initiated on inhaled treprostinil sodium for treatment of PAH who have concomitant COPD.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2011-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in Oxygen saturation in subject initiated on inhaled treprostinil sodium for treatment of PAH who have concomintant COPD. | Dec 2014

SECONDARY OUTCOMES:
Change in 6MWT in subject initiated on inhaled treprostinil sodium for treatment of PAH who have concomintant COPD. | December 2014

OTHER OUTCOMES:
SGRQ questionaires | December 2014

CONTACTS AND LOCATIONS:
Overall Officials: Abubakr A Bajwa, MD, FCCP, Principal Investigator — University of Florida
Locations (3):
- United States (3):
  - University of Florida, Jacksonville, Jacksonville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Cleveland Clinic Florida, Weston, Florida